CLINICAL TRIAL: NCT01772576
Title: RELIANCE 4-FRONT™ Active Fixation Defibrillation Lead Post Market Clinical Follow-Up (PMCF) Study
Brief Title: Safety and Performance Study of the Reliance 4-Front Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSC-CDM00052753; C1830 (Other Grant/Funding Number: C1830)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2016-04

CONDITIONS: Tachycardia
Keywords: Reliance; Implantable Cardioverter Defibrillator (ICD); Cardiac Resynchronization Therapy - Defibrillator (CRT-D)
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Reliance 4-Front (Experimental): Single arm, all patients will be implanted with the Reliance 4-Front lead
  Interventions: Device: Reliance 4-Front lead implantation

INTERVENTIONS:
Device: Reliance 4-Front lead implantation — The patients selected for participation should be from the investigator's general patient population with an indication for implantation of a single or dual chamber ICD or CRT-D system.

SUMMARY:
The objective of this study is to gather data to establish the chronic safety, performance and effectiveness of the RELIANCE 4-FRONT™ Active Fixation Defibrillation Leads.

DETAILED DESCRIPTION:
The RELIANCE 4-FRONT Defibrillation Lead Post Market Clinical Follow-Up Study is a prospective, non-randomized, multi-center, single-group, post market clinical study to establish the chronic safety, performance and effectiveness of the RELIANCE 4-FRONT active fixation defibrillation leads.

A total of 167 patients (including 10 % attrition) are required to evaluate the Primary Endpoint.

Up to 20 Investigational centers located in Europe and Asia Pacific. Lead-related Complication-Free Rate (CFR) from Implant through 3 Months Post-Implant.

Lead-related complications associated with the RELIANCE 4-FRONT active fixation lead will count toward this endpoint.

Lead-related Complication-Free Rate from 3 Months through 15 Months Post-Implant.

Lead-related complications associated with the RELIANCE 4-FRONT active fixation lead will count toward this endpoint.

* Lead-related Complication-Free Rate from 3 Months through 24 Months Post-Implant
* Pacing Threshold at 0.5 ms pulse width at 3 Months Post-Implant
* Sensed Amplitude at 3 Months Post-Implant
* Pacing Impedance at 3 Months Post-Implant All endpoints will be assessed for the RELIANCE 4-FRONT active fixation lead.

Clinic visits will occur at:

* Enrollment Visit (no later than 30 days prior to implant procedure)
* Implant Procedure (Day 0; all future follow ups based on this date)
* Pre-Discharge Clinic Visit (3 - 72 hours post-implant)
* One Month Clinic Visit (30±7 days)
* 3 Month Clinic Visit (91 ± 21 days)
* 6 Month Clinic Visit (180 ± 30 days)
* 12 Month Clinic Visit (365 ± 45 days)
* 18 Month Clinic Visit (545± 45 days)
* 24 Month Clinic Visit (730 ± 45 days) The study will be considered completed after all subjects have completed the 24 Month follow-up and study completion is anticipated in 2015. Primary endpoint completion is anticipated after all subjects have completed the 3 Month follow-up visit. All study required visits will be completed during clinic visits.

Hypotheses testing in the RELIANCE 4-FRONT PMCF Study will use standard statistical methodology as specified more in detail in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of providing informed consent
* Has an indication for implantation of a single or dual chamber ICD or CRT-D system in their respective geography
* Subjects planned to be implanted with the RELIANCE 4-FRONT Active Fixation Lead
* Willing and capable of participating in all testing/ visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
* Age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Known or suspected sensitivity to Dexamethasone Acetate (DXA)
* Mechanical tricuspid heart valve
* Subject is enrolled in any other concurrent study without prior written approval from Boston Scientific (BSC), with the exception of local mandatory governmental registries and observational studies/registries that are not in conflict and do not affect the following:
* Schedule of procedures for the RELIANCE 4-Front Study (i.e. should not cause additional or missed visits);
* RELIANCE 4-Front Study outcome (i.e. involve medications that could affect the heart rate of the subject);
* Conduct of the RELIANCE 4-Front Study per Good Clinical Practice (GCP)/ International Organization for Standardization (ISO) 14155:2011/ 21 CFR 812/ local regulations
* Currently on the active heart transplant list
* Documented life expectancy of less than 12 months
* Women of childbearing potential who are or might be pregnant at the time of study enrollment (method of assessment upon physician discretion)
* Currently requiring chronic dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Bongiorni, MD, Principal Investigator — University Hospital Pisa, Italy
Locations (15):
- Landesklinikum St. Poelten, Sankt Pölten, Austria
- Queen Mary Hospital, Hong Kong, China
- Aarhus University Hospitals, Aarhus, Denmark
- Institut Cardiovasculaire - Paris Sud, Massy, France
- Germany (2):
  - Deutsches Herzzentrum Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
- Israel (2):
  - Barzilai Medical Center, Ashkelon
  - Sheba Medical Center, Tel Litwinsky
- Italy (2):
  - Ospedale Alessandro Manzoni, Lecco
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Hospital de Santa Cruz, Carnaxide, Portugal
- Hospital Universitario Virgen de la Victoria, Málaga, Spain
- Karolinska Hospital, Stockholm, Sweden
- United Kingdom (2):
  - Bristol Royal Infirmary, Bristol
  - Golden Jubilee National Hospital, Clydebank

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 167 patients were enrolled in the study. Patients were considered enrolled when the consent form was signed regardless whether they received the RELIANCE 4FRONT lead or not. Recruitment started on 22 November 2012. Last patient was enrolled 9 March 2014.
Pre-assignment Details: No wash out or run-in period was planned for the study. 3 patients did not receive the study lead: lead not available at site, wrong lead chosen and patient needed MRI (magnet resonance imaging) compatible lead, while the RELIANCE 4FRONT lead was not labeled MRI compatible.
Groups:
- Reliance 4-Front: Single arm, all patients were implanted with the Reliance 4-Front lead
  Reliance 4-Front lead implantation: The patients selected for participation were from the investigator's general patient population with an indication for implantation of a single or dual chamber ICD or CRT-D system.
Period: Overall Study
Arm/Group | Reliance 4-Front
Started | 167
Completed | 133
Not Completed | 34
Not completed — Death | 15
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 3
Not completed — Study device not used | 3
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Reliance 4-Front
Number analyzed (Participants) | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.26 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 138
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 10
  Sweden | 9
  China | 10
  Denmark | 25
  United Kingdom | 22
  Italy | 15
  Israel | 44
  France | 4
  Portugal | 4
  Germany | 20
  Spain | 4

OUTCOME MEASURES:

1. Primary Outcome: Complication Free Rate
Description: Lead-related Complication-Free Rate (CFR) from Implant through 3 Months Post-Implant.
Time Frame: 3-months follow-up
Population: Patients enrolled in the study and having received the RELIANCE 4FRONT active fixation lead
Measure: Number (95% Confidence Interval); unit: percentage of all subjects
Arm/Group | Reliance 4-Front
Number analyzed (Participants) | 164
percentage of all subjects | 96.3 [92.9 to 99.7]

2. Secondary Outcome: Complication Free Rate
Description: Lead-related Complication-Free Rate from 3 Months through 15 Months Post-Implant.
Time Frame: 3 months through 15 months post implant
Population: 156 patients remained after 3 months in the study without lead related complication. Those were used for the secondary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of total participants
Arm/Group | Reliance 4-Front
Number analyzed (Participants) | 156
percentage of total participants | 98.7 [95.8 to 100]

3. Other Pre Specified Outcome: Complication Free Rate
Description: Lead-related Complication-Free Rate from 3 Months through 24 Months Post-Implant
Time Frame: 3 Months through 24 Months Post-Implant
Population: Patients remaining after the 3 months follow-up in the study until the 24 months follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of all participants
Arm/Group | Reliance 4-Front
Number analyzed (Participants) | 156
percentage of all participants | 98.7 [95.8 to 100]

4. Other Pre Specified Outcome: Pacing Threshold
Description: Pacing Threshold at 0.5 ms pulse width at 3 Months Post-Implant
Time Frame: 3-months post-implant
Population: Patients having undergone the 3 months follow-up visit.
Measure: Mean (95% Confidence Interval); unit: Volt
Arm/Group | Reliance 4-Front
Number analyzed (Participants) | 144
Volt | 0.53 [0.48 to 0.58]

5. Other Pre Specified Outcome: Sensed Amplitude
Description: Sensed Amplitude at 3 Months Post-Implant
Time Frame: 3 Months Post-Implant
Population: Patients having undergone the 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: mV
Arm/Group | Reliance 4-Front
Number analyzed (Participants) | 144
mV | 18.1 [17.1 to 19.1]

6. Other Pre Specified Outcome: Pacing Impedance
Description: Pacing Impedance at 3 Months Post-Implant
Time Frame: 3 Months Post-Implant
Population: Patients with 3 month follow-up
Measure: Mean (95% Confidence Interval); unit: Ohm
Arm/Group | Reliance 4-Front
Number analyzed (Participants) | 150
Ohm | 474 [457 to 491]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through 24 months.
Description: Definitions do not differ from clinicaltrials.gov definitions
Arm/Group | Reliance 4-Front
All-Cause Mortality (participants affected / at risk) | 14/164
Serious Adverse Events (participants affected / at risk) | 89/167
Other Adverse Events (participants affected / at risk) | 69/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Reliance 4-Front (N=167)
Inappropriate tachy therapy - SVT (Cardiac disorders) | 1/164 (1)
Inappropriate tachy therapy - Other (Cardiac disorders) | 1/164 (1)
Erosion (Skin and subcutaneous tissue disorders) | 1/164 (1)
Infection (> 30 days post-implant) (Infections and infestations) | 3/164 (3)
Psychological effect due to device therapy (Psychiatric disorders) | 2/164 (2)
Post-surgical wound discomfort (Skin and subcutaneous tissue disorders) | 1/164 (1)
Post-surgical pocket hemorrhage (Skin and subcutaneous tissue disorders) | 1/164 (1)
Adverse reaction - General (General disorders) | 1/164 (1)
Hemorrhage (Injury, poisoning and procedural complications) | 1/164 (1)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 2/164 (2)
Unable to capture - RV (General disorders) | 2/164 (2)
Elevated threshold - RV (General disorders) | 1/164 (1)
Impedance > 2000 ohms - RV (General disorders) | 2/164 (2)
Dislodgment - Multiple signs - RV (General disorders) | 1/164 (1)
Dislodgment - No reported signs - RV (General disorders) | 1/164 (1)
Elevated threshold - LV (General disorders) | 1/164 (1)
Dislodgment - Elevated threshold - LV (General disorders) | 1/164 (1)
Dislodgment - No reported signs - LV (General disorders) | 1/164 (1)
Pneumothorax - Procedure (Injury, poisoning and procedural complications) | 1/164 (1)
Coronary venous dissection (Vascular disorders) | 1/164 (1)
Other - Lead - Procedure: implant failure (General disorders) | 1/164 (1)
Pulseless electrical activity (PEA) (Cardiac disorders) | 1 (1)
VENTRICULAR TACHYARRHYTHMIAS (Cardiac disorders) | 1 (1)
Ventricular fibrillation (VF) (Cardiac disorders) | 4 (5)
Ventricular tachycardia (VT) (Cardiac disorders) | 5 (9)
Torsades des pointes (Cardiac disorders) | 2 (2)
Atrial fibrillation (AF) (Cardiac disorders) | 9 (14)
Atrial flutter (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Premature ventricular contractions (PVC) (Cardiac disorders) | 1 (1)
Syncope - Heart failure (Cardiac disorders) | 3 (3)
Chest pain - Heart failure (Cardiac disorders) | 2 (2)
Dyspnea - Heart failure (Cardiac disorders) | 5 (5)
Peripheral edema - Heart failure (Cardiac disorders) | 1 (1)
Pulmonary edema - Heart failure (Cardiac disorders) | 3 (7)
Fatigue - Heart failure (Cardiac disorders) | 1 (1)
Dehydration - Heart failure (Cardiac disorders) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 4 (4)
Multiple heart failure symptoms (Cardiac disorders) | 9 (12)
Multi-system failure - Heart failure (Cardiac disorders) | 8 (8)
Coronary Artery Disease (Vascular disorders) | 3 (3)
Peripheral vascular disease (Vascular disorders) | 3 (4)
Syncope (Vascular disorders) | 6 (6)
Chest pain - Ischemic (Cardiac disorders) | 2 (3)
Chest pain - Other (Cardiac disorders) | 6 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Multiple symptoms (General disorders) | 2 (2)
Cerebrovascular accident (CVA) (Vascular disorders) | 4 (4)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Death (General disorders) | 4 (4)
Systemic infection (Infections and infestations) | 1 (1)
Fever (General disorders) | 1 (1)
Physical trauma (Injury, poisoning and procedural complications) | 1 (1)
Abnormal laboratory values (Blood and lymphatic system disorders) | 1 (2)
Hematological (Blood and lymphatic system disorders) | 5 (8)
Neurological (Nervous system disorders) | 2 (3)
Gastrointestinal (Gastrointestinal disorders) | 11 (16)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Genitourinary (Renal and urinary disorders) | 4 (7)
Renal (Renal and urinary disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4)
Psychological (Psychiatric disorders) | 1 (1)
Integumentary (Skin and subcutaneous tissue disorders) | 2 (2)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1 (1)
Endocrine (Endocrine disorders) | 3 (3)
Cancer (General disorders) | 5 (6)
Multi-system failure (General disorders) | 1 (1)
Adverse drug reaction (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Reliance 4-Front (N=167)
Unable to capture - RA (Cardiac disorders) | 1/164 (1)
Inappropriate tachy therapy - Other (Cardiac disorders) | 1/164 (2)
Post-surgical wound discomfort (Skin and subcutaneous tissue disorders) | 1/164 (2)
Post-surgical infection (<= 30 days post-implant) (Skin and subcutaneous tissue disorders) | 3/164 (3)
Adverse reaction - General (General disorders) | 3 (3)
Adverse reaction - Respiratory (Respiratory, thoracic and mediastinal disorders) | 1/164 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1/164 (1)
Hematoma - Pocket (<=30 days post-implant) (Injury, poisoning and procedural complications) | 8/164 (8)
Other-PG system-Procedure: Other non system related (Injury, poisoning and procedural complications) | 1/164 (1)
Dislodgment - Multiple signs - RV (General disorders) | 1/164 (1)
Unable to capture - LV (General disorders) | 1/164 (1)
Elevated threshold - LV (General disorders) | 3/164 (3)
Extracardiac stimulation - LV (General disorders) | 4/164 (5)
Dislodgment - Elevated threshold - LV (General disorders) | 1/164 (1)
Pneumothorax - Procedure (Injury, poisoning and procedural complications) | 1/164 (1)
Other - Lead - Procedure: difficulties due to venous access (General disorders) | 1/164 (1)
wound infection after LV lead placement (Infections and infestations) | 1/164 (1)
Ventricular tachycardia (VT) (Cardiac disorders) | 5 (5)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 3 (3)
ATRIAL TACHYARRHYTHMIAS (Cardiac disorders) | 2 (2)
Atrial fibrillation (AF) (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Other SVT (AVRT, AVNRT, EAT etc.) (Cardiac disorders) | 1 (1)
Dyspnea - Heart failure (Cardiac disorders) | 7 (8)
Peripheral edema - Heart failure (Cardiac disorders) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Syncope (Vascular disorders) | 1 (3)
Dizziness (General disorders) | 2 (2)
Chest pain - Other (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Deep vein thrombosis (DVT) (Vascular disorders) | 1 (1)
Localized infection (Infections and infestations) | 1 (1)
Physical trauma (Injury, poisoning and procedural complications) | 7 (7)
Hematological (Blood and lymphatic system disorders) | 1 (1)
Neurological (Nervous system disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Genitourinary (Renal and urinary disorders) | 5 (5)
Renal (Renal and urinary disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (6)
Psychological (Psychiatric disorders) | 3 (3)
Integumentary (Skin and subcutaneous tissue disorders) | 3 (3)
Head, eyes, ears, nose, throat (HEENT) (Infections and infestations) | 2 (2)
Endocrine (Endocrine disorders) | 4 (4)
Immune (Immune system disorders) | 1 (1)
Cancer (Blood and lymphatic system disorders) | 1 (1)
Adverse drug reaction (General disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Sample size was rather small and power of the study is only 80%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes